CLINICAL TRIAL: NCT00150410
Title: A One-Year, Open, Randomized, Parallel, Three-Arm Study Comparing Exubera® (Insulin Dry Powder Pulmonary Inhaler) vs. Avandia® (Rosiglitazone Maleate) as Add-On Therapy vs. Exubera® Substitution of Sulfonylurea in Patients With Type 2 Diabetes, Poorly Controlled on Combination Sulfonylurea and Metformin Treatment
Brief Title: Demonstrate Exubera Works As Well As Avandia When Added To Sulfonylurea + Metformin In Controlling Glucose
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A2171017
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2008-10-31 (Estimated); Status verified 2008-10

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

INTERVENTIONS:
Drug: Inhaled insulin

SUMMARY:
* Whether a combination of three therapies - metformin and a sulfonylurea plus Exubera, an investigational drug, controls your diabetes at least as much as a triple combination therapy of metformin and a sulfonylurea plus Avandia, a Food and Drug Administration (FDA) approved drug.
* Whether a combination of two therapies - metformin plus Exubera controls your diabetes at least as much as a as a triple combination therapy of metformin and a sulfonylurea plus Avandia.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Currently treated and on a stable doses of drugs for the preceding two (2) months

Exclusion Criteria:

* Type 1 Diabetes
* Smoking

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 626 (Actual)
Dates: Start 2003-01; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Glycosylated hemoglobin

SECONDARY OUTCOMES:
Change from baseline in fasting plasma glucose. Other secondary efficacy
endpoints include, body weight, patient reported outcomes, incidence and severity
of hypoglycemic episodes, cough questionnaire, and discontinuation rate due to
insufficient clinical response.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (101):
- United States (75):
  - Pfizer Investigational Site, Mesa, Arizona
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Searcy, Arkansas
  - Pfizer Investigational Site, Alhambra, California
  - Pfizer Investigational Site, Concord, California
  - Pfizer Investigational Site, Huntington Beach, California
  - Pfizer Investigational Site, La Jolla, California
  - Pfizer Investigational Site, Long Beach, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Riverside, California
  - Pfizer Investigational Site, Santa Barbara, California
  - Pfizer Investigational Site, Tustin, California
  - Pfizer Investigational Site, Westminster, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Wheat Ridge, Colorado
  - Pfizer Investigational Site, Waterbury, Connecticut
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Hollywood, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Winter Park, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Augusta, Georgia
  - Pfizer Investigational Site, Savannah, Georgia
  - Pfizer Investigational Site, Honolulu, Hawaii
  - Pfizer Investigational Site, ‘Ewa Beach, Hawaii
  - Pfizer Investigational Site, Idaho Falls, Idaho
  - Pfizer Investigational Site, Chicago Heights, Illinois
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Des Moines, Iowa
  - Pfizer Investigational Site, Wichita, Kansas
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Baton Rouge, Louisiana
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Springfield, Massachusetts
  - Pfizer Investigational Site, Waltham, Massachusetts
  - Pfizer Investigational Site, West Saint Paul, Minnesota
  - Pfizer Investigational Site, North Kansas City, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Butte, Montana
  - Pfizer Investigational Site, Lincoln, Nebraska
  - Pfizer Investigational Site, New Brunswick, New Jersey
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, Albany, New York
  - Pfizer Investigational Site, Flushing, New York
  - Pfizer Investigational Site, Mineola, New York
  - Pfizer Investigational Site, New Hyde Park, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Lakewood, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Duncan, South Carolina
  - Pfizer Investigational Site, Spartanburg, South Carolina
  - Pfizer Investigational Site, Sumter, South Carolina
  - Pfizer Investigational Site, Kingsport, Tennessee
  - Pfizer Investigational Site, Knoxville, Tennessee
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Corpus Christi, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, El Paso, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Ogden, Utah
  - Pfizer Investigational Site, Fredericksburg, Virginia
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Renton, Washington
  - Pfizer Investigational Site, Tukwila, Washington
  - Pfizer Investigational Site, Milwaukee, Wisconsin
- Australia (7):
  - Pfizer Investigational Site, Camperdown, New South Wales
  - Pfizer Investigational Site, Wollongong, New South Wales
  - Pfizer Investigational Site, Herston, Queensland
  - Pfizer Investigational Site, Woolloongabba, Queensland
  - Pfizer Investigational Site, Keswick, South Australia
  - Pfizer Investigational Site, Box Hill, Victoria
  - Pfizer Investigational Site, Caulfield, Victoria
- Brazil (2):
  - Pfizer Investigational Site, Porto Alegre, Rio Grande do Sul
  - Pfizer Investigational Site, São Paulo, São Paulo
- Canada (11):
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Mississauga, Ontario
  - Pfizer Investigational Site, Oakville, Ontario
  - Pfizer Investigational Site, Thornhill, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Laval, Quebec
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Saint-Jérôme, Quebec
  - Pfizer Investigational Site, Vaudreuil, Quebec
  - Pfizer Investigational Site, St. John's
- Mexico (6):
  - Pfizer Investigational Site, Guadalajara, Jalisco
  - Pfizer Investigational Site, Guadalajara, Jalisco/Mexico
  - Pfizer Investigational Site, Mexico City, Mexico City
  - Pfizer Investigational Site, Monterrey, Nuevo León
  - Pfizer Investigational Site, Jalapa, Veracruz
  - Pfizer Investigational Site, Mexico City

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2171017&StudyName=Demonstrate%20Exubera%20Works%20As%20Well%20As%20Avandia%20When%20Added%20To%20Sulfonylurea%20+%20Metformin%20In%20Controlling%20Glucose